CLINICAL TRIAL: NCT01029925
Title: A Multicenter, Phase II Open-Labeled, Single-Arm Clinical and Pharmacology Study of Dichloroacetate (DCA) in Patients With Previously Treated Metastatic Breast or Non-Small Cell Lung Cancer
Brief Title: Dichloroacetate (DCA) in Patients With Previously Treated Metastatic Breast or Non-Small Cell Lung Cancer (NSCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB determined, due to higher than expected risk/safety concerns, study should be closed.
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCA Breast NSCLC; 09-07-013 (Other: UCLA IRB)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2013-06

CONDITIONS: Metastatic Breast Cancer; Lung Cancer
Keywords: metastatic breast cancer; lung cancer; Previously treated metastatic breast cancer; stage IIIb lung cancer; stage IV lung cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms | interventions — Dichloroacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dichloroacetate (DCA) (Experimental): Dichloroacetate, 6.25mg/kg orally, twice daily, administered with food around the same time every day and at approximately 8-12 hours apart.
  Interventions: Drug: Dichloroacetate (DCA)

INTERVENTIONS:
Drug: Dichloroacetate (DCA) — Dichloroacetate, 6.25mg/kg orally, twice daily, administered with food around the same time every day and at approximately 8-12 hours apart

SUMMARY:
The purpose of this study is to determine the response rate by RECIST criteria of oral dichloroacetate in patients with recurrent and/or metastatic and pretreated breast and non-small cell lung cancer.

DETAILED DESCRIPTION:
In the United States, approximately 180,000 new cases of breast cancer occur annually, and there are more than 40,000 deaths. More than 150,000 cases develop each year in Canada and the European community together, resulting in over 60,000 deaths from breast cancer. The vast majority of patients who die from breast cancer succumb to metastatic disease. Endocrine therapy and chemotherapy (using either sequential single agents or combination regimens) remain the principal treatments for women with metastatic breast cancer. A wide variety of classes of chemotherapeutic agents have activity as single agents. Median survival remains approximately two years for women with metastatic breast cancer, and less than 3% of patients will experience long-term survival after treatment. The development of new treatment strategies is therefore essential to improve outcome for patients with metastatic breast cancer. The population selected for this study will have previously received, where appropriate, those drugs with clearly defined survival advantages (anthracyclines, taxanes, trastuzumab, and hormonal therapy).

Patients with metastatic non-small cell lung cancer are considered incurable. Palliative chemotherapies, such as platinum-based doublet, Taxotere or Pemetrexed or Erlotinib (an epidermal growth factor tyrosine kinase) have been proven to improve symptoms, and survival in patients with good performance status. Despite these treatments, the median survival of metastatic non-small cell lung cancer is about one year. Therefore, there is an urgent need to develop novel therapy in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic breast cancer or Stage IIIb or IV non-small cell lung cancer.
* Must have measurable disease as defined by at least one target lesion by RECIST criteria that has not been irradiated.
* Progressive disease after prior chemotherapy or patient refusal of these chemotherapy options.

  * Breast Cancer

    * Patients should have received two prior lines of chemotherapy. This should include prior anthracycline and taxane therapy, either in the adjuvant or metastatic setting.
    * HER-2 positive breast cancer should have received Trastuzumab, in either the adjuvant or metastatic setting.
    * Estrogen Receptor positive breast cancer should have received at least one prior hormonal therapy, either in the adjuvant or metastatic setting.
  * Non-small cell lung cancer patients should have received at least platinum based chemotherapy in the adjuvant, neoadjuvant or metastatic setting.
* Age > 18 years.
* ECOG performance status < 2.
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count >1,500/mcL
  * Hemoglobin >9.0 g/dL
  * Platelets >100,000/mcL
  * Total bilirubin <1.5 X upper limit of normal (ULN)
  * AST (SGOT) and ALT (SGPT) <2.5 X ULN or <5 X ULN in the presence of live metastases.
  * Creatinine <1.5 X ULN
* Recovery to baseline or, at most, grade 1 of all drug-related toxicities due to prior chemotherapy, radiation, hormonal therapy, or molecular targeted therapy, except for alopecia.
* Ejection fraction by MUGA scan or echocardiogram must be within normal range.
* Women of childbearing potential must have a negative pregnancy test and women and men must agree to use adequate contraception prior to study entry, for the duration of study participation and for 30 days after the last dose of study therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy, hormonal therapy, molecular targeted therapy, or radiotherapy within 4 weeks prior to receiving first dose of DCA. An exception will be made for palliative radiation to bone which must have been completed 10 days prior to the first dose of DCA. An exception will also be made for HER-2 positive BC who can continue to receive Trastuzumab during therapy with DCA.
* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents, chemotherapy, immunotherapy, radiotherapy, or molecular targeted agents.
* Active CNS metastasis.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to DCA.
* Due to the possibility of peripheral sensorimotor neuropathy from DCA, the presence of any grad peripheral neuropathy due to prior medical condition (such as multiple sclerosis), medications, or other etiologies.
* Any psychological, familial, sociological, or geographical conditions that do not permit medical follow-up and compliance with the study protocol.
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection (requiring parenteral anti-biotics), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with DCA.
* 2 years must have elapsed since the initial curative procedure for other malignancies, except for in situ cervical cancer, non-melanoma skin cancer, and localized prostate cancer after curative therapy such as surgery, or radiation.
* Patient history of inflammatory bowel disease, malabsorption syndrome, condition causing chronic diarrhea and requiring active therapy or substantial amount of small bowels or stomach removed that may impair absorption of DCA.
* Therapeutic anticoagulation will be allowed with Heparin or LMWH but not with Coumadin.
* Any history of nephrolithiasis because of possible increase in urinary oxalate with DCA and correlation with nephrolithiasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garon, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Kjaer A. Molecular imaging of cancer using PET and SPECT. Adv Exp Med Biol. 2006;587:277-84. PMID 17163171
- [Background] Warburg O. Ueber den stoffweschsel der tumoren (London: Constable). (1930).
- [Background] Gatenby RA, Gillies RJ. Why do cancers have high aerobic glycolysis? Nat Rev Cancer. 2004 Nov;4(11):891-9. doi: 10.1038/nrc1478. PMID 15516961
- [Background] Merida I, Avila-Flores A. Tumor metabolism: new opportunities for cancer therapy. Clin Transl Oncol. 2006 Oct;8(10):711-6. doi: 10.1007/s12094-006-0117-6. PMID 17074669
- [Background] Andersson B, Janson V, Behnam-Motlagh P, Henriksson R, Grankvist K. Induction of apoptosis by intracellular potassium ion depletion: using the fluorescent dye PBFI in a 96-well plate method in cultured lung cancer cells. Toxicol In Vitro. 2006 Sep;20(6):986-94. doi: 10.1016/j.tiv.2005.12.013. Epub 2006 Feb 17. PMID 16483738
- [Background] Remillard CV, Yuan JX. Activation of K+ channels: an essential pathway in programmed cell death. Am J Physiol Lung Cell Mol Physiol. 2004 Jan;286(1):L49-67. doi: 10.1152/ajplung.00041.2003. PMID 14656699
- [Background] Wang H, Zhang Y, Cao L, Han H, Wang J, Yang B, Nattel S, Wang Z. HERG K+ channel, a regulator of tumor cell apoptosis and proliferation. Cancer Res. 2002 Sep 1;62(17):4843-8. PMID 12208728
- [Background] Yu SP, Yeh CH, Sensi SL, Gwag BJ, Canzoniero LM, Farhangrazi ZS, Ying HS, Tian M, Dugan LL, Choi DW. Mediation of neuronal apoptosis by enhancement of outward potassium current. Science. 1997 Oct 3;278(5335):114-7. doi: 10.1126/science.278.5335.114. PMID 9311914
- [Background] Bonnet S, Archer SL, Allalunis-Turner J, Haromy A, Beaulieu C, Thompson R, Lee CT, Lopaschuk GD, Puttagunta L, Bonnet S, Harry G, Hashimoto K, Porter CJ, Andrade MA, Thebaud B, Michelakis ED. A mitochondria-K+ channel axis is suppressed in cancer and its normalization promotes apoptosis and inhibits cancer growth. Cancer Cell. 2007 Jan;11(1):37-51. doi: 10.1016/j.ccr.2006.10.020. PMID 17222789
- [Derived] Garon EB, Christofk HR, Hosmer W, Britten CD, Bahng A, Crabtree MJ, Hong CS, Kamranpour N, Pitts S, Kabbinavar F, Patel C, von Euw E, Black A, Michelakis ED, Dubinett SM, Slamon DJ. Dichloroacetate should be considered with platinum-based chemotherapy in hypoxic tumors rather than as a single agent in advanced non-small cell lung cancer. J Cancer Res Clin Oncol. 2014 Mar;140(3):443-52. doi: 10.1007/s00432-014-1583-9. Epub 2014 Jan 18. PMID 24442098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with breast cancer (1) and non-small cell lung cancer (6) were recruited at UCLA between January 2010 and December 2010.
Pre-assignment Details: One patient developed a brain metastasis before beginning therapy and had to be excluded, and two patients were undergoing screening procedures when the study was placed on voluntary hold.
Period: Completion of Cycle 1 (28 Days)
Arm/Group | Dichloroacetate (DCA)
Started | 7
Completed | 3
Not Completed | 4
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Period: Completion of Cycle 2 (56 Days)
Arm/Group | Dichloroacetate (DCA)
Started | 3
Completed | 2
Not Completed | 1
Not completed — off study due to disease progression | 1

BASELINE CHARACTERISTICS:
Population: Stage 1 has best prognosis and stage IV has worst.Grade 1 is associated with best prognosis and grade 3 with poor prognosis.ECOG performance status grades a person's overall well-being and scaled from 0-5.ECOG of 0 is associated with best prognosis.Patients with ECOG 0-2 are considered well enough to receive additional treatments for their cancer.
Arm/Group | Dichloroacetate (DCA)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
stage at diagnosis [Number; unit: participants]
  Stage II breast cancer | 1
  Stage IV NSCLC | 6
ECOG status [Number; unit: participants]
  ECOG status 0 | 2
  ECOG status 1 | 3
  ECOG status 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Response Rate by RECIST Criteria of Oral Dichloroacetate in Patients With Recurrent and/or Metastatic and Pretreated Breast and Non-small Cell Lung Cancer.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: upto 72 days
Population: Intent to treat analysis was performed. Zero patients achieved complete or partial response in this study.
Measure: Number; unit: participants
Arm/Group | Dichloroacetate (DCA)
Number analyzed (Participants) | 7
participants | 0

ADVERSE EVENTS:
Arm/Group | Dichloroacetate (DCA)
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dichloroacetate (DCA) (N=7)
Sudden death (General disorders) | 2 (2)
pulmonary embolism (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dichloroacetate (DCA) (N=7)
abdominal pain (Gastrointestinal disorders) | 2 (3)
Fever (General disorders) | 1 (1)
fatigue (General disorders) | 2 (3)
lower extremity edema (Blood and lymphatic system disorders) | 2 (3)
urinary retention (Renal and urinary disorders) | 1 (1)
Dyspnea (General disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 1 (1)
Xerostomia (General disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
tremor (General disorders) | 1 (1)
nausea (General disorders) | 1 (1)
candidiasis (Infections and infestations) | 2 (2)
disequilibrium (General disorders) | 2 (2)
lower extremity coldness (General disorders) | 1 (1)
elevated AST (Metabolism and nutrition disorders) | 1 (1)
pain (General disorders) | 2 (2)
seizures (General disorders) | 1 (1)
hyponatremia (General disorders) | 1 (1)
volume depletion (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The greatest limitation in our study was early termination due to perceived lack of drug efficacy leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No